CLINICAL TRIAL: NCT01121029
Title: Autologous Hematopoietic Stem Cell Transplantation in Type 1 Diabetes Mellitus
Brief Title: Hematopoietic Stem Cell Transplantation in Type 1 Diabetes Mellitus
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Dra. Olga Graciela Cantu Rodriguez (Other)
Responsible Party: Sponsor-Investigator, Dra. Olga Graciela Cantu Rodriguez, Autologous Hematopoietic Stem Cell Transplantation in Type 1 Diabetes Mellitus, Hospital Universitario Dr. Jose E. Gonzalez
Organization: Hospital Universitario Dr. Jose E. Gonzalez (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EN10-011
Record Dates: First submitted 2010-05-11; First posted 2010-05-12 (Estimated); Last update posted 2012-12-10 (Estimated); Status verified 2012-12

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Hematopoietic stem cells (Experimental)
  Interventions: Procedure: Autologous hematopoietic stem cell transplantation

INTERVENTIONS:
Procedure: Autologous hematopoietic stem cell transplantation — Patients will receive a stimulation with filgrastim 10mcg/Kg per day during 4 days and cyclophosphamide 1.5g/m2 per day during 2 days and mesna 300mg/m2 i.v. in 4 hours for prophylaxis (uroprotection). Lately, the stem cells will be recollected by apheresis. After that, the patients will receive a conditioning regimen with cyclophosphamide 500mg/m2 per day during 4 days and fludarabine 30mg/m2 per day during 4 days. After the last dose of cyclophosphamide, the autologous hematopoietic stem cell transplantation will be done on day 0, by peripheral vein. Then, a standard regimen of prophylaxis with oral ciprofloxacin 500mg every 12 hours, acyclovir 400mg every 8 hours, fluconazole 100mg per day and omeprazole 20mg per day for the recovery time of each patient.
  Other Names: Stem cell therapy

SUMMARY:
The purpose of this study is to determine if autologous nonmyeloablative hematopoietic stem cell transplantation is able to induce prolonged and significant increases of C-peptide levels associated with absence of or reduction of daily insulin.

DETAILED DESCRIPTION:
Patients with type 1 DM depend on exogenous insulin administration for survival and for control of long-term complications. The best-established treatment is tight control of blood glucose achieved by frequent daily injections or continuous subcutaneous infusion of insulin, ie, intensive insulin therapy. Although insulin therapy has developed enormously, even the most modern technologies do not allow the maintenance of normoglycemia.

Since the establishment of the autoimmune etiology of type 1 DM in the late 1970s, many clinical trials analyzing the effects of different types of immune interventions demonstrated that beta-cell preservation is an achievable target in different degrees.

Controlled trials and further biological studies are necessary to confirm the role of this treatment in changing the natural history of type 1 DM.

This is a prospective pilot study which will enroll patients with type 1 diabetes mellitus within the first months of diagnosis, with clinical and laboratory findings. The donor stimulation will be with cyclophosphamide, filgrastim, and mesna. The cells will be recollected from peripheral blood by apheresis and refrigerated. The patients will receive a nonmyeloablative conditioning regimen with cyclophosphamide and fludarabine, and after this, the cells will be injected intravenously. They will receive a standard regimen of post-transplant prophylaxis. The duration of use of this prophylactic drugs scheme depends on the patient's recovery time. The reinfusion of stem cells will be completed after the last dose of cyclophosphamide, through a peripheral vein.

Lately, every three months, the C-Peptide levels, glucose and insulin serum levels will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed in type 1 diabetes mellitus

Exclusion Criteria:

* Patients with HIV
* Patients with Hepatitis
* Patients with hematologic disease
* Patients with hearth failure
* Renal, Hepatic or psychiatric disease
* Pregnant patients

Ages: 2 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2010-05; Primary Completion 2011-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
C-peptide levels before and after the hematopoietic stem cell transplantation | Every 3 months for 1 year.

SECONDARY OUTCOMES:
Serum levels of Hb A1C before and after the hematopoietic stem cell transplantation | Every month for 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Fernando J Lavalle, MD, Principal Investigator — Hospital Universitario Dr. José Eleuterio González; David Gómez, MD, Study Chair — Hospital Universitario Dr. José Eleuterio González; Olga G Cantú, MD, Study Director — Hospital Universitario Dr. José Eleuterio González
Locations (1):
- Hospital Universitario Dr. José Eleuterio González, Monterrey, Nuevo León, Mexico

REFERENCES:
- [Background] Couri CE, Voltarelli JC. Potential role of stem cell therapy in type 1 diabetes mellitus. Arq Bras Endocrinol Metabol. 2008 Mar;52(2):407-15. doi: 10.1590/s0004-27302008000200029. PMID 18438552
- [Background] Couri CE, Foss MC, Voltarelli JC. Secondary prevention of type 1 diabetes mellitus: stopping immune destruction and promoting beta-cell regeneration. Braz J Med Biol Res. 2006 Oct;39(10):1271-80. doi: 10.1590/s0100-879x2006001000002. Epub 2006 Aug 22. PMID 16941054
- [Background] Voltarelli JC, Couri CE, Stracieri AB, Oliveira MC, Moraes DA, Pieroni F, Coutinho M, Malmegrim KC, Foss-Freitas MC, Simoes BP, Foss MC, Squiers E, Burt RK. Autologous nonmyeloablative hematopoietic stem cell transplantation in newly diagnosed type 1 diabetes mellitus. JAMA. 2007 Apr 11;297(14):1568-76. doi: 10.1001/jama.297.14.1568. PMID 17426276
- [Background] Voltarelli JC, Couri CE. Stem cell transplantation for type 1 diabetes mellitus. Diabetol Metab Syndr. 2009 Sep 16;1(1):4. doi: 10.1186/1758-5996-1-4. PMID 19825196
- [Background] Effect of intensive therapy on residual beta-cell function in patients with type 1 diabetes in the diabetes control and complications trial. A randomized, controlled trial. The Diabetes Control and Complications Trial Research Group. Ann Intern Med. 1998 Apr 1;128(7):517-23. doi: 10.7326/0003-4819-128-7-199804010-00001. PMID 9518395
- [Background] Couri CE, Oliveira MC, Stracieri AB, Moraes DA, Pieroni F, Barros GM, Madeira MI, Malmegrim KC, Foss-Freitas MC, Simoes BP, Martinez EZ, Foss MC, Burt RK, Voltarelli JC. C-peptide levels and insulin independence following autologous nonmyeloablative hematopoietic stem cell transplantation in newly diagnosed type 1 diabetes mellitus. JAMA. 2009 Apr 15;301(15):1573-9. doi: 10.1001/jama.2009.470. PMID 19366777
- [Result] Otonkoski T, Gao R, Lundin K. Stem cells in the treatment of diabetes. Ann Med. 2005;37(7):513-20. doi: 10.1080/07853890500300279. PMID 16278164
- [Derived] Cantu-Rodriguez OG, Lavalle-Gonzalez F, Herrera-Rojas MA, Jaime-Perez JC, Hawing-Zarate JA, Gutierrez-Aguirre CH, Mancias-Guerra C, Gonzalez-Llano O, Zapata-Garrido A, Villarreal-Perez JZ, Gomez-Almaguer D. Long-Term Insulin Independence in Type 1 Diabetes Mellitus Using a Simplified Autologous Stem Cell Transplant. J Clin Endocrinol Metab. 2016 May;101(5):2141-8. doi: 10.1210/jc.2015-2776. Epub 2016 Feb 9. PMID 26859103